CLINICAL TRIAL: NCT07373002
Title: Development, Optimization, and Effectiveness Evaluation of an Intelligent Parent-Infant Connection-Based Family Resilience Intervention: A Longitudinal Study of Parental Psychosocial Health From Hospitalization to Post-Discharge in Preterm Infants
Brief Title: Development and Evaluation of an Intelligent Parent-Infant Connection-Based Intervention to Strengthen Family Resilience in Preterm Infant Care
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Defense Medical Center, Taiwan (Other)
Responsible Party: Principal Investigator, Hsiang-Yun Lan, Associate Professor, National Defense Medical Center, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: T-NDMU-67611
Record Dates: First submitted 2026-01-13; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Family Resilience; Parent-Infant Bonding; Parents of Premature Infants; Intelligent Intervention
Keywords: Psychosocial Health; Digital Health Intervention; Salivary Cortisol; Neonatal Intensive Care Unit (NICU); Physical Health; Social Health; Mental Health; Family Resilience; Parent-Infant Bonding
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intelligent Intervention to enhance Parent-Infant Connection and Family Resilience (Experimental): Participants in this group will receive routine care plus an intelligent parent-infant connection-based intervention. The intervention includes access to a mobile platform that delivers structured educational content focused on premature infant care, emotional regulation, parent-infant bonding, and stress management. The program begins during the infant's NICU hospitalization and continues for one month post-discharge. Participants will also receive interactive messages, tips, and guidance to support their caregiving role and psychosocial adjustment during the transition to home care.
  Interventions: Behavioral: Intelligent Intervention to enhance Parent-Infant Connection and Family Resilience; Other: Routine Care
- Routine care group (Active Comparator): Participants in this group will receive routine care as provided in the NICU and after discharge, including standard parent education and support without access to the digital intervention program. They will complete the same assessments as the experimental group across five time points from hospitalization to six months post-discharge.
  Interventions: Other: Routine Care

INTERVENTIONS:
Behavioral: Intelligent Intervention to enhance Parent-Infant Connection and Family Resilience — This is a structured, mobile-based behavioral intervention designed to support the psychosocial health and caregiving competence of parents with preterm infants during and after NICU hospitalization. The intervention includes educational modules, interactive messages, and self-guided activities delivered through a digital platform. Content is tailored to promote parent-infant bonding, enhance parenting confidence, strengthen family resilience, and reduce parenting stress. The intervention begins during the infant's NICU stay and continues for one month after discharge. Participants receive reminders, feedback, and supportive information based on their responses and needs, aiming to facilitate the transition from hospital to home and improve early parenting experiences.
  Arms: Intelligent Intervention to enhance Parent-Infant Connection and Family Resilience
Other: Routine Care — Participants in this group will receive routine care as provided in the NICU and after discharge, including standard parent education and support without access to the digital intervention program. They will complete the same assessments as the experimental group across five time points from hospitalization to six months post-discharge.

SUMMARY:
This study aims to develop, optimize, and evaluate the effectiveness of a family resilience intervention centered on intelligent parent-infant connection for parents of preterm infants. Using a longitudinal randomized controlled trial design, it examines the intervention's impact on parental psychosocial health, parenting efficacy, family resilience, and parent-infant interaction from NICU hospitalization to six months post-discharge.

DETAILED DESCRIPTION:
This longitudinal randomized controlled trial evaluates a family resilience intervention centered on intelligent parent-infant connection, designed for parents of preterm infants hospitalized in the NICU. The study recruits approximately 150 dyads of preterm infants' parents over three years at Tri-Service General Hospital, Taiwan. The intervention group receives routine care plus a digitally delivered support program during hospitalization and the first month after discharge, while the control group receives routine clinical care only. The intervention comprises low-burden, accessible modules focusing on parent-infant interaction, caregiving competence, emotional support, and paternal involvement. Data are collected at five time points: baseline (within 1 week of NICU admission), pre-discharge, and one, three, and six months post-discharge. Outcomes include family resilience, parenting efficacy, parent-infant bonding, psychological stress, sleep quality, and biological stress indicators (salivary cortisol). The study aims to establish the intervention's effectiveness in improving the psychosocial well-being of preterm infants' parents and supporting family adaptation across care transitions.

ELIGIBILITY:
Inclusion Criteria:

* The infant is born prematurely with a gestational age of less than 37 weeks.
* At least one parent of the premature infant is aged 18 years or older and can communicate in Mandarin or Taiwanese.
* The parent(s) have provided informed consent to participate in the study.
* The parent(s) are able to comply with the data collection procedures (participation of both parents is encouraged but not required).

Exclusion Criteria:

* The premature infant has major congenital anomalies or is assessed by clinicians as unlikely to survive.
* The parent(s) are unable to use a smartphone or internet-connected device due to technical, cognitive, or other limitations.
* The parent(s) have a known history of severe psychiatric disorders, intellectual disabilities, or substance abuse, and are assessed by the research team as being unable to comply with the study procedures or intervention requirements.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in Family Resilience | At baseline (before intervention), 1 month after birth, and at 1 month, 3 months, and 6 months post-discharge.
  Family resilience will be measured using the Chinese version of the Walsh Family Resilience Questionnaire. This scale assesses key processes across three domains: family belief systems, organizational patterns, and communication/problem-solving. Each item is rated on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). The total score is calculated by summing item scores, with higher scores indicating greater family resilience.
Change in Parent-Infant Bonding | At baseline (before intervention), 1 month after birth, and at 1 month, 3 months, and 6 months post-discharge.
  Parent-infant bonding will be assessed using the Chinese version of the Postpartum Bonding Questionnaire (PBQ), which measures the parent's emotional connection to their infant, including feelings of affection, confidence, and potential rejection or anxiety. The scale includes 25 items rated on a 6-point scale from 0 (always) to 5 (never), with some items reverse scored. Total scores range from 0 to 125; lower scores indicate stronger parent-infant bonding, while higher scores suggest bonding difficulties.
Change in Perceived Stress | At baseline (before intervention), 1 month after birth, and at 1 month, 3 months, and 6 months post-discharge.
  Perceived stress will be measured using the Chinese version of the 14-item Perceived Stress Scale (PSS-14). This scale assesses participants' subjective evaluation of stress in their lives during the past month. Each item is rated on a 5-point Likert scale from 0 (never) to 4 (very often). The total score ranges from 0 to 56, with higher scores indicating higher levels of perceived stress.
Change in Postpartum Specific Anxiety | At baseline (before intervention), 1 month after birth, and at 1 month, 3 months, and 6 months post-discharge.
  Postpartum anxiety will be measured using the Chinese version of the Postpartum Specific Anxiety Scale - Research Short Form (PSAS-RSF-C). The scale includes 16 items evaluating anxiety related to infant care, maternal competence, psychosocial adjustment, and infant safety. Items are rated on a 4-point Likert scale from 1 (not at all) to 4 (very much). Total scores range from 16 to 64, with higher scores indicating greater postpartum-specific anxiety.
Change in Salivary Cortisol | At baseline (before intervention), 1 month after birth, and at 1 month, 3 months, and 6 months post-discharge.
  Cortisol levels (in ng/mL) serve as a physiological biomarker for stress; higher levels indicate greater stress reactivity. Salivary cortisol levels will be collected using a non-invasive saliva collection method and analyzed using the SOMA real-time cortisol analysis system. Saliva samples will be collected at consistent times to control for diurnal variation.
Change in Family Hardiness | At baseline (before intervention), 1 month after birth, and at 1 month, 3 months, and 6 months post-discharge.
  The Family Hardiness Index (FHI) assesses family resilience in response to stress and crisis. It consists of 20 items measuring three dimensions: commitment, control, and challenge. Each item is rated on a 4-point Likert scale ranging from 1 (strongly disagree) to 4 (strongly agree), with items 1, 2, 3, 8, 10, 14, 16, 19, and 20 reverse scored. Total scores range from 20 to 80, with higher scores indicating greater family hardiness and stronger coping abilities.
Change in Maternal Postnatal Attachment | At baseline (before intervention), 1 month after birth, and at 1 month, 3 months, and 6 months post-discharge.
  The Maternal Postnatal Attachment Scale (MPAS) evaluates the emotional quality of maternal attachment to the infant. It includes 19 items across three dimensions: quality of attachment, absence of hostility, and pleasure in interaction. Each item is re-coded to a uniform 5-point scale from 1 to 5, with some items reverse scored. Total scores range from 19 to 95, with higher scores reflecting stronger and more positive maternal attachment.
Change in Maternal Confidence | At baseline (before intervention), 1 month after birth, and at 1 month, 3 months, and 6 months post-discharge.
  The Maternal Confidence Questionnaire assesses a mother's perceived confidence in parenting, particularly in the context of premature infants. The scale consists of 14 items rated on a 5-point Likert scale from 1 (never) to 5 (always), with items 12 and 14 reverse scored. Higher total scores indicate greater maternal confidence.
Change in Parental Role Adaptation | At baseline (before intervention), 1 month after birth, and at 1 month, 3 months, and 6 months post-discharge.
  The Parental Role Adaptation Scale in Neonatal Intensive Care Units assesses mothers' adaptation to the maternal role during their infant's NICU stay. It consists of 32 items rated on a 5-point Likert scale from 1 (strongly disagree) to 5 (strongly agree), covering six domains: involvement in care (14 items), self-efficacy (6), remote motherhood (3), uncertainty (4), interaction (3), and growth and development (2). Higher scores indicate better adaptation to the maternal role.
Change in Functional Social Support | At baseline (before intervention), 1 month after birth, and at 1 month, 3 months, and 6 months post-discharge.
  The Functional Social Support Scale measures caregivers' perceived social support across three dimensions: support needed, assistance received, and satisfaction. Each of the 16 items includes aspects of emotional, informational, and instrumental support. Responses are given on a 5-point Likert scale ranging from 0 (never) to 4 (always), or from 0 (not needed at all) to 4 (very much needed). Higher scores indicate stronger perceived support and fulfillment.

SECONDARY OUTCOMES:
Change in Quality of Life | At baseline (before intervention), 1 month after birth, and at 1 month, 3 months, and 6 months post-discharge.
  Measured using the Taiwan version of WHOQOL-BREF, which contains 26 items covering physical, psychological, social, and environmental domains. Each item is rated on a 5-point scale. Total scores are calculated and standardized to a 0-100 scale, with higher scores indicating better quality of life.
Change in Parental Self-Efficacy | At baseline (before intervention), 1 month after birth, and at 1 month, 3 months, and 6 months post-discharge.
  Parental self-efficacy will be assessed using the Parental Self-Efficacy Scale (PSE), a 20-item instrument scored on a 5-point Likert scale from 1 (strongly disagree) to 5 (strongly agree). Scores range from 20 to 100. Higher scores indicate stronger parental confidence in caregiving roles.
Change in Subjective Sleep Quality | At baseline (before intervention), 1 month after birth, and at 1 month, 3 months, and 6 months post-discharge.
  Evaluated using the Pittsburgh Sleep Quality Index (PSQI), which includes 19 items assessing sleep duration, latency, quality, and disturbances. Scores range from 0 to 21, with higher scores indicating worse sleep quality. A score >5 suggests poor sleep.
Change in Objective Sleep Indicators | At baseline (before intervention), 1 month after birth, and at 1 month, 3 months, and 6 months post-discharge.
  Sleep duration and efficiency will be measured using the ActiGraph GT3X accelerometer, worn continuously on the non-dominant wrist for 72 hours. Data will be downloaded and analyzed to calculate total sleep time (minutes) and sleep efficiency (percentage of time asleep while in bed).
Change in Subjective Sleep Quality and Parameter (Sleep Diary) | At baseline (before intervention),1 month after birth, and at 1 month, 3 months, and 6 months post-discharge.
  This self-developed sleep diary was designed to capture sleep quality, patterns, and disturbances over a continuous 3-day period. Each morning upon waking, participants recorded their recall of the previous night's sleep, including total sleep time (in hours), number and duration of nighttime awakenings, and perceived sleep efficiency. They also noted contextual factors that may have affected their sleep, such as emotional distress, physical discomfort, medication use, or consumption of stimulants or alcohol. In addition, participants rated their perceived sleep quality and level of alertness upon waking using a 5-point Likert scale, where 1 indicated the poorest quality or alertness and 5 indicated the highest. Higher scores reflect better subjective sleep outcomes.

IPD SHARING:
Plan to Share IPD: No